CLINICAL TRIAL: NCT04047212
Title: Analysis of the Link Between Periodontitis, Smoking and Oral Cancer: Cohort Study
Brief Title: The Link Between Periodontitis, Smoking and Oral Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayat Gamal-AbdelNaser, Principal investigator, Cairo University
Other Study IDs: P12
Record Dates: First submitted 2019-08-03; First posted 2019-08-06 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Chronic Periodontitis; Oral Cancer
MeSH Terms: conditions — Chronic Periodontitis; Mouth Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — biopsy of cases having oral lesions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokers
  Interventions: Diagnostic Test: biopsy for oral cancer; Diagnostic Test: periodontal examination
- non-Smokers
  Interventions: Diagnostic Test: biopsy for oral cancer; Diagnostic Test: periodontal examination

INTERVENTIONS:
Diagnostic Test: biopsy for oral cancer — surgical biopsy is to be taken for diagnosis of oral cancer or premalignant lesions
Diagnostic Test: periodontal examination — Periodontal clinical examination to all by periodontal charting

SUMMARY:
Periodontitis is a widely prevalent disease worldwide that has serious public health consequences. Its prognosis includes tooth loss and edentulism, a condition that negatively affects chewing causing functional disability; and esthetics causing social impairment. Consequently, periodontitis may end up causing marked impairment of the quality of life of the affected patients, impairment of general health and increasing the dental care costs significantly.

Changes in the oral mucosa arise by primary products resulting from tissue breakdown due to gingivitis. It then triggers the host cells to produce proteinases that mediate loss of marginal periodontal ligaments, apical migration of the junctional epithelium and apical spread of bacterial biofilm.

Therefore, this research aims to identify the risk of smoking to both periodontitis and oral cancer, and the risk of periodontitis to oral cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.

Exclusion Criteria:

* Patients with any systemic diseases.
* Pregnant females.
* Handicapped and mentally retarded patients.
* Patients undergoing radiotherapy.
* Patients having oral cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult individuals
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-08-12 (Estimated); Primary Completion 2031-10-12 (Estimated); Study Completion 2032-01-30 (Estimated)

PRIMARY OUTCOMES:
Periodontitis | the 10 years of the study
  arising of periodontitis or increase in the grade of an already existing case of periodontitis

SECONDARY OUTCOMES:
Oral cancer | the 10 years of the study
  Arising of a lesion of oral cancer or a premalignant lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No